CLINICAL TRIAL: NCT03625362
Title: Effects of Hydrogen-rich Water on Liver Fat Accumulation, Blood Lipids and Body Fatness in Patients With Non-alchoholic Fatty Liver Disease
Brief Title: Hydrogen-rich Water for Non-alchoholic Fatty Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Novi Sad, Faculty of Sport and Physical Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 0417-HRW/2018
Record Dates: First submitted 2018-08-06; First posted 2018-08-10 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Hydrogen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrogen (Experimental): 1 L of hydrogen-rich water
  Interventions: Dietary Supplement: Hydrogen
- Placebo (Placebo Comparator): 1 L of tap water
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Hydrogen — Hydrogen-rich water
  Arms: Hydrogen
Dietary Supplement: Placebo — Tap water
  Arms: Placebo

SUMMARY:
This study evaluates how 4-week supplementation with hydrogen-rich water affects liver fat accumulation, blood lipid profiles and body composition in patients with non-alcoholic fatty liver disease

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is a metabolic disorder characterized by liver fat deposition due to causes other than excessive alcohol consumption. NAFLD can cause many liver dysfunction-related symptoms and signs, with the disease may progress to non-alcoholic steatohepatitis, a condition marked by liver inflammation, fibrosis and irreversible damage. NAFLD is usually accompanied by insulin resistance and obesity, with up to 30% of population in industrialized countries have NAFLD. While NAFLD is rapidly becoming the most common liver disease worldwide, its treatment remains elusive, and directed toward correction of the risk factors. Since metabolic impairment plays a major role in NAFLD pathogenesis, any agent that advance lipid and glucose metabolism could be appropriate to tackle this complex condition. Molecular hydrogen (H2) has recently emerged as a novel pro-metabolic agent that might positively affect liver health. Supplemental hydrogen improves blood lipid profiles and insulin resistance in overweight women, patients with type 2 diabetes, and in subjects with potential metabolic syndrome. In addition, drinking hydrogen-rich water reduces hepatic oxidative stress and alleviated fatty liver damage in rodents. However, no human studies so far evaluated its effectiveness to alter liver steatosis in patients with NAFLD. In this pilot trial, we analyze the effects of 4-week hydrogen-rich water intake on liver fat deposition, body composition and lab chemistry profiles in overweight patients suffering from NAFLD.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Body mass index > 25 kg/m2
* Free of major diseases besides NAFLD
* Must be able to give written informed consent

Exclusion Criteria:

* Use of any dietary supplements within 4 weeks before study commences
* Abnormal values for lab clinical chemistry (> 2 SD)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Liver fat content | Change from baseline liver triglycerides at 4 weeks
  MRS spectra for liver triglycerides

SECONDARY OUTCOMES:
Total cholesterol | Change from baseline total cholesterol at 4 weeks
  Level of total cholesterol in the blood
Total body fatness | Change from baseline fat percentage at 4 weeks
  Fat percentage evaluated by BIA

CONTACTS AND LOCATIONS:
Locations (2):
- Serbia (2):
  - Applied Bioenergetics Lab at Faculty of Sport and PE, Novi Sad, Vojvodina
  - FSPE Applied Bioenergetics Lab, Novi Sad, Vojvodina

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared via Institutional repository

REFERENCES:
- [Background] Kajiyama S, Hasegawa G, Asano M, Hosoda H, Fukui M, Nakamura N, Kitawaki J, Imai S, Nakano K, Ohta M, Adachi T, Obayashi H, Yoshikawa T. Supplementation of hydrogen-rich water improves lipid and glucose metabolism in patients with type 2 diabetes or impaired glucose tolerance. Nutr Res. 2008 Mar;28(3):137-43. doi: 10.1016/j.nutres.2008.01.008. PMID 19083400
- [Background] Nakao A, Toyoda Y, Sharma P, Evans M, Guthrie N. Effectiveness of hydrogen rich water on antioxidant status of subjects with potential metabolic syndrome-an open label pilot study. J Clin Biochem Nutr. 2010 Mar;46(2):140-9. doi: 10.3164/jcbn.09-100. Epub 2010 Feb 24. PMID 20216947
- [Background] Korovljev D, Trivic T, Drid P, Ostojic SM. Molecular hydrogen affects body composition, metabolic profiles, and mitochondrial function in middle-aged overweight women. Ir J Med Sci. 2018 Feb;187(1):85-89. doi: 10.1007/s11845-017-1638-4. Epub 2017 May 30. PMID 28560519
- [Derived] Korovljev D, Stajer V, Ostojic J, LeBaron TW, Ostojic SM. Hydrogen-rich water reduces liver fat accumulation and improves liver enzyme profiles in patients with non-alcoholic fatty liver disease: a randomized controlled pilot trial. Clin Res Hepatol Gastroenterol. 2019 Nov;43(6):688-693. doi: 10.1016/j.clinre.2019.03.008. Epub 2019 Apr 11. PMID 30982748